CLINICAL TRIAL: NCT05612308
Title: Effects of Vertical Oscillatory Pressure and Sustained Natural Apophyseal Glides on Pain- Biomakers, Selected Clinical and Psychosocial Variables in Patients With Mechanical Low- Back -Pain
Brief Title: Vertical Oscillatory Pressure and Sustained Natural Apophyseal Glides in ow Back Pain
Acronym: VOP&SNAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Obafemi Awolowo University (Other)
Responsible Party: Principal Investigator, Adesola Ojo Ojoawo, Principal Investigator, Obafemi Awolowo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ojo/2022/02
Record Dates: First submitted 2022-10-31; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Non Specific Low Back Pain
Keywords: Low back pain,; Vertical Oscillatory Pressure,; Sustained Natural Apophzeal Glide,; Pain-Biomakers; Health Related Quality of Life
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: There were two groups; Vertical Oscillatory and Sustained Natural Apophyseal group. Participants were allocated to each group randomly. Each group received intervention accordingly
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verical Oscillatory Pressure (VOP) (Experimental): Vertical Oscillatory Pressure (VOP) will be administered with the patient lying prone on a couch. The researcher will place the thumb reinforced with the other thumb on the implicated lumbar vertebra, then apply pressure posterior anteriorly on the spinous process and oscillate for a maximum of 60 seconds. This will be done on each patient in this group twice a week for 6 weeks after an initial assessment both subjective and objective (Egwu et al, 2007).
  Interventions: Other: Vertical Oscillatory Pressure (VOP)
- Sustained Natural Apophyzeal Glides (Experimental): Participant in this group will undergo SNAG technique on lumbar vertebra with active spinal movement according to Mulligan, (2004). Participants will be in a sitting position on the edge of the couch while both feet will be on a footrest. A stabilization belt will be used around the patient's waist and the therapist's hips and the researcher standing behind the patient well supported with stabilization belt. The researcher places one thumb or hypothenar eminence (pisiform bone) reinforced by the other on the spinous process of the implicated lumbar vertebra and then apply pressure posterior-anteriorly on the spinous process, the pressure will be sustained and the patient concurrently performs active spinal movement. SNAGS will be applied with 3 repetitions on the first day and 10 repetitions from next visit. SNAG will be used twice a week for 6 weeks.
  Interventions: Other: Vertical Oscillatory Pressure (VOP)

INTERVENTIONS:
Other: Vertical Oscillatory Pressure (VOP) — The VOP involves a pressure from the posterior aspect of the body while patient lye prone. the pressure is exacted directly on the spine, The sustained Natural Apophyseal Glides involves pressure as well when the patient sits down on a chair. The movement is done from the posterior to the anterior as well
  Other Names: Sustained Natural Apophyseal Glides (SNAGs)

SUMMARY:
Among different spinal manual therapies, which have been reported to be effective in the management of LBP are Sustained Natural Apophyseal Glide (SNAGS) and Vertical Oscillatory Pressure (VOP) . Vertical oscillatory pressure is a derivative of manipulative therapy whereby a gentle vertical manipulative oscillation is applied on spinal vertebrae and has been noted to be effective in management of low back pain . On the contrary, the SNAGS is a manipulative technique that is commonly used in the western countries and found to be effective in reducing pain and disability in the management of mechanical LBP . However, there are limited studies comparing the effects of SNAG and VOP on clinical and psychosocial variables in patients with mechanical LBP in Nigeria. Hence, this study aims at investigating the effects of Nwugarian VOP and SNAG techniques on selected clinical and psychosocial variables in patients with mechanical LBP.

DETAILED DESCRIPTION:
Low back pain and the attendant disabilities have been on the increase in Africa and its burden is more in countries with longer life expectancy . The menace of the condition includes high level of disability, producing significant restrictions on usual activity and participation, such as ability to work . Contrary to general belief, LBP is not a problem that always resolves by itself, recurrences are usual and the course is varying in different circumstances . While emerging evidence and advocacy by Physiotherapy Associations favours active treatment for long-term LBP, however, spinal manipulation remains an important option for LBP that will or not resolve with active and self-care. Spinal manipulation has been reported to produce significant benefits within a short period , may be more and faster than expected improvements with active therapies . Further, while there is increasing advocacy for active management of LBP, many patients are not well suited or positioned to treat themselves, hence may require experts' management.

Sustained Natural Apophyseal Glide (SNAGS) is a manipulative technique that is commonly used in the western countries and found to be effective in reducing pain and disability in the management of mechanical LBP . In another study by Shabana et al., on the comparative effect of SNAGS and Maitland's mobilization in chronic LBP, better improvement was observed in SNAGS group than in Maitland's. however, it is not commonly used in the Nigerian context. On the other hand, the Nwugarian technique; VOP, propunded by Nwuga is a home-grown spinal manipulation approach in Nigeria demonstrated the effectiveness of VOP on pain and disability in patients with mechanical lowback pain. VOP, in combination with lumbar stabilization exercises has also been noted to be more effective compared with VOP in isolation in the management chronic low back pain . Similarly, Egwu et al., concluded that VOP has significant effects on pain intensity and Lumbo-sacral mobility, and opined that VOP should be preferred as spinal mobilization therapy outcome measures in youths and elderly individuals with LBP. The effectiveness of VOP is hinged on few available studies. VOP requires pressure on the vertebral spinous process with oscillation by the therapist. The therapeutic mechanism of spinal manipulation have emphasized the importance of directing forces to specific spinal joints for the purpose of correcting a biomechanical dysfunction or misalignment . Studies have also shown and validated spinal manipulation to affect both sensory and motor nerve activity as well as electromyographic measured muscle activity . Outcome measures reflect the impact of the health care service or intervention on the health status of patients. To achieve comprehensive multidimensional evaluation of outcome in LBP ,one of the core outcome domains that must be considered is pain, the method of assessing has always been participants rating of improvement and satisfaction with treatment but not the effects of intervention at cellular level. Use of serum biomarkers has the potential to measure the effects of intervention at cellular level thereby helping to identify relevant treatment options and decrease the likelihood of failed interventions. However, effects of known treatment like VOP and SNAGS on the inflammatory status and bio cellular pain substance in patients with long term low-back pain has not been explored, ,hence this study This study is therefore aimed to investigate and compare the effect of VOP and SNAGS on pain-biomarkers, disability, flexibility and health-related quality of life in patients with mechanical LBP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non specific low back pain of at least 3 months duration
* age of 18-75 years
* No history of hospitalization in the last 12 months

Exclusion Criteria:

* No history of trauma
* organic diseases
* No mental disorderliness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 6 weeks
  Pain perception: Which is measured by Visual Analogue Scale . This is an instrument that measure the pain perception of the patients. The minimum is 0, which indicated no pain and the maximum is 10 which described excruciating pain

SECONDARY OUTCOMES:
Interleuking 6 | 6 weeks
  Concentration of pain factors in the blood. It is an chemical in the blood that determines how individuals perceive pain in the body. The minimum is 30 which indicate no pain and the maximum could be 250 which indicate extreme pain

CONTACTS AND LOCATIONS:
Overall Officials: Adesola O Ojoawo, PhD, Principal Investigator — Obafemi Awolowo University Ile ife
Locations (1):
- Obafemi Awolowo University, Ile-Ife, Osun State, Nigeria

IPD SHARING:
Plan to Share IPD: No
The data may not be shared with other researchers

REFERENCES:
- [Background] Ojoawo AO, Olaogun MO, Odejide SA, Badru AA. Effect of vertical oscillatory pressure on disability of patients with chronic mechanical low back pain using Roland Morris Disability questionnaire. Tanzan J Health Res. 2013 Jan;15(1):58-63. doi: 10.4314/thrb.v15i1.9. PMID 26591674
- [Background] Ogunlana MO, Odole AC, Adejumo A, Odunaiya N. Catastrophising, pain, and disability in patients with nonspecific low back pain. Hong Kong Physiother J. 2015 Dec;33(2):73-79. doi: 10.1016/j.hkpj.2015.03.001. Epub 2015 Apr 16. PMID 30930571
- [Background] Roche RJ, Silamut K, Pukrittayakamee S, Looareesuwan S, Molunto P, Boonamrung S, White NJ. Quinine induces reversible high-tone hearing loss. Br J Clin Pharmacol. 1990 Jun;29(6):780-2. doi: 10.1111/j.1365-2125.1990.tb03704.x. PMID 2198912